CLINICAL TRIAL: NCT01371981
Title: A Phase III Randomized Trial for Patients With De Novo AML Using Bortezomib and Sorafenib (NSC# 681239, NSC# 724772) for Patients With High Allelic Ratio FLT3/ITD
Brief Title: Bortezomib and Sorafenib Tosylate in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02670; NCI-2011-02670 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000701850; AAML1031; COG-AAML1031; S12-02301; AAML1031 (Other: Children's Oncology Group); AAML1031 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Leukemia Cutis; Myeloid Neoplasm; Myeloid Sarcoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Sarcoma, Myeloid | interventions — Asparaginase; Leyk; Bortezomib; Cytarabine; Daunorubicin; Etoposide; Mitoxantrone; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (6):
- Arm A (Experimental): See Detailed Description
  Interventions: Drug: Asparaginase; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (Experimental): See Detailed Description
  Interventions: Drug: Asparaginase; Drug: Bortezomib; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm C (Cohort 1) (Experimental): See Detailed Description
  Interventions: Drug: Asparaginase; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sorafenib Tosylate
- Arm C (Cohort 2) (Experimental): See Detailed Description.
  Interventions: Drug: Asparaginase; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sorafenib Tosylate
- Arm C (Cohort 3) (Experimental): See Detailed Description. Different dose.
  Interventions: Drug: Asparaginase; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sorafenib Tosylate
- Arm D (Experimental): See Detailed Description. May reassigned to Arm C.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Asparaginase — Given IM
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-Asparaginase; L-Asparagine Amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa; Spectrila
  Arms: Arm A; Arm B; Arm C (Cohort 1); Arm C (Cohort 2); Arm C (Cohort 3)
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; LDP-341; LDP341; MLN 341; MLN-341; MLN341; PS 341; PS-341; PS341; Velcade
  Arms: Arm B
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
  Arms: Arm A; Arm B; Arm C (Cohort 1); Arm C (Cohort 2); Arm C (Cohort 3)
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54 9085; BAY 54-9085; BAY 549085; BAY-54-9085; BAY549085; Nexavar; sorafenib
  Arms: Arm C (Cohort 1); Arm C (Cohort 2); Arm C (Cohort 3)

SUMMARY:
This randomized phase III trial studies how well bortezomib and sorafenib tosylate work in treating patients with newly diagnosed acute myeloid leukemia. Bortezomib and sorafenib tosylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib and sorafenib tosylate together with combination chemotherapy may be an effective treatment for acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare event-free survival (EFS) and overall survival (OS) in patients with de novo acute myeloid leukemia (AML) without high allelic ratio fms-like tyrosine kinase (FLT3)/internal tandem duplications (ITD)+ mutations who are randomized to standard therapy versus bortezomib/standard combination therapy.

II. To determine the feasibility of combining bortezomib with standard chemotherapy in patients with de novo AML.

III. To compare the OS and EFS of high-risk patients treated with intensive Induction II with historical controls from AAML03P1 and AAML0531.

IV. To determine the feasibility of administering sorafenib (sorafenib tosylate) with standard chemotherapy and in a one year maintenance phase in patients with de novo high allelic ratio FLT3/ITD+ AML.

SECONDARY OBJECTIVES:

I. To assess the anti-leukemic activity of sorafenib in patients with de novo high allelic ratio FLT3/ITD+ AML.

II. To compare the percentage of patients converting from positive minimal residual disease (MRD) to negative MRD after Intensive Induction II with historical controls from AAML03P1 and AAML0531.

III. To compare OS, disease-free survival (DFS), cumulative incidence of relapse, and treatment-related mortality from end of Intensification I between patients allocated to best allogenic donor stem cell transplant (SCT) and comparable patients on AAML0531 who did not receive allogenic donor SCT.

IV. To compare OS, DFS, cumulative incidence of relapse, treatment-related mortality, and severe toxicity between patients allocated to matched family donor SCT on AAML1031 and AAML0531.

V. To assess the health-related quality of life (HRQOL) of patients treated with chemotherapy and stem cell transplant (SCT) for AML.

VI. To evaluate bortezomib pharmacokinetics (PK) in patients receiving the combination regimen.

VII. To obtain sorafenib and metabolite steady state pharmacokinetics and pharmacokinetic-pharmacodynamic data in subjects with FLT3/ITD receiving sorafenib.

VIII. To compare the changes in shortening fraction/ejection fraction over time between patients treated with and without dexrazoxane.

IX. To refine the use of minimal-residual disease (MRD) detection with 4-color flow cytometry.

X. To evaluate the prognostic significance of molecular MRD and its contribution to risk identification with multidimensional flow cytometry (MDF)-based MRD in patients with translocations amenable to quantitative real time (RT)-polymerase chain reaction (PCR) (e.g., t[8;21], inv[16], t[9;11], Wilms tumor 1 [WT1] expression).

XI. To determine the leukemic involvement of the hematopoietic early progenitor cell and its role in defining response to therapy.

XII. To define the leukemic stem cell population in patients with AML. XIII. To determine the prevalence and prognostic significance of molecular abnormalities of WT1, runt-related transcription factor (RUNX)1, mixed-lineage leukemia (MLL)-partial tandem duplication (PTD), tet methylcytosine dioxygenase 2 (TET2), Cbl proto-oncogene, E3 ubiquitin protein ligase (c-CBL), v-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (KIT), and other novel AML-associated genes in pediatric AML.

XIV. Correlate the expression of cluster of differentiation (CD)74 antigen as well as proteasome beta 5-subunit (PSMB5) gene expression and mutation with response to bortezomib.

XV. To evaluate the changes in protein expression and unfolded protein response (UPR) in patients with AML.

XVI. To determine the expression level of wild-type FLT3, and correlate with outcome and in vitro sensitivity to FLT3 inhibition.

XVII. To collect biology specimens at diagnosis, treatment time points, and relapse for future biology studies XVIII. To create a pediatric-specific algorithm to predict the occurrence of grade 2-4 acute graft-versus-host disease (GVHD) prior to its clinical manifestations using a combination of pre-transplant clinical variables and serum GVHD biomarker concentrations in the first weeks after SCT.

OUTLINE: This is a dose-escalation study of sorafenib tosylate. Patients are randomized to Arm A or B or offered treatment on 1 of 6 arms. (Arms A and B are closed to new patient enrollment as of 02/04/2016)

Arm A:

INDUCTION I: Patients receive cytarabine intrathecally (IT) on day 1 and ADE chemotherapy comprising cytarabine intravenously (IV) over 1-30 minutes on days 1-10; daunorubicin hydrochloride IV over 1-15 minutes on days 1, 3, and 5; and etoposide IV over 1-2 hours on days 1-5.

INDUCTION II: Patients with low risk (LR) receive cytarabine IT and ADE chemotherapy as in Induction I. Patients with high risk (HR) receive cytarabine IT on day 1 and MA chemotherapy comprising high-dose cytarabine IV over 1-3 hours on days 1-4, and mitoxantrone IV over 15-30 minutes on days 3-6. Patients who achieve complete remission (CR) proceed to Intensification I (beginning on day 37). Patients with refractory disease are off protocol therapy.

INTENSIFICATION I: Patients receive cytarabine IT on day 1 and AE chemotherapy comprising high-dose cytarabine IV over 1-3 hours, and etoposide IV over 1-2 hours on days 1-5. Patients who achieve CR proceed to Intensification II or stem cell transplantation (SCT) beginning on day 34. Patients with refractory disease are off protocol therapy.

INTENSIFICATION II: Patients with LR receive cytarabine IT on day 1 and MA chemotherapy as in Induction II. Patients with HR and no donor for SCT receive high-dose cytarabine IV over 3 hours on days 1, 2, 8, and 9 and asparaginase intramuscularly (IM) on days 2 and 9.

STEM CELL TRANSPLANTATION (SCT) (HR patients with matched family [MFD] or unrelated donor):

CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily on days -5 to -2.

TRANSPLANTATION: Patients undergo allogeneic SCT within 36 to 48 hours after the last dose of busulfan.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or PO beginning on day -2 and continuing until day 98 (matched sibling donor) or day 180 (with taper) (other related/unrelated donors or cord blood) and methotrexate IV on days 1, 3, and 6 (matched sibling/cord blood donors) or days 1, 3, 6, and 11 (other related/unrelated donors). Patients with unrelated donors also receive antithymocyte globulin IV over 6-8 hours on days -3 to -1.

Arm B:

INDUCTION I: Patients receive cytarabine IT and ADE chemotherapy as in Induction I, Arm A. Patients also receive bortezomib IV over 3-5 seconds on days 1, 4, and 8.

INDUCTION II: Patients with LR receive cytarabine IT, ADE chemotherapy, and bortezomib as in Induction I. Patients with HR receive cytarabine IT and MA chemotherapy as in Induction II, Arm A (HR patients) and bortezomib IV on days 1, 4, and 8.

INTENSIFICATION I: Patients receive cytarabine IT and AE chemotherapy in Arm A, Intensification II, and bortezomib IV on days 1, 4, and 8. Patients who achieve CR proceed to Intensification II or stem cell transplantation (SCT) beginning on day 34. Patients with refractory disease are off protocol therapy.

INTENSIFICATION II: Patients with LR receive cytarabine IT on day 1, MA chemotherapy as in Arm A, Induction II (HR patients), and bortezomib IV on days 1, 4, and 8. Patients with HR and no donor for SCT receive high-dose cytarabine IV over 3 hours on days 1, 2, 8, and 9 and asparaginase intramuscularly (IM) on days 2 and 9.

STEM CELL TRANSPLANTATION (SCT) (HR patients with matched family [MFD] or unrelated donor):

CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily on days -5 to -2.

TRANSPLANTATION: Patients undergo allogeneic SCT within 36 to 48 hours after the last dose of busulfan.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or PO beginning on day -2 and continuing until day 98 (matched sibling donor) or day 180 (with taper) (other related/unrelated donors or cord blood) and methotrexate IV on days 1, 3, and 6 (matched sibling/cord blood donors) or days 1, 3, 6, and 11 (other related/unrelated donors). Patients with unrelated donors also receive antithymocyte globulin IV over 6-8 hours on days -3 to -1.

ARM C (COHORT 1):

INDUCTION II: Patients receive cytarabine IT on day 1, cytarabine IV over 1-30 minutes on days 1-8, daunorubicin hydrochloride IV over 1-15 minutes on days 1, 3, and 5, etoposide IV over 1-2 hours on days 1-5, and sorafenib tosylate PO on days 9-36.

INTENSIFICATION I: Patients receive cytarabine IT and AE chemotherapy in Arm A, Intensification II, and sorafenib tosylate PO on daily on days 6-28.

INTENSIFICATION II: Patients receive cytarabine IT on day 1, MA chemotherapy as in Arm A, Induction II (HR patients), and sorafenib tosylate PO on days 7-34.

STEM CELL TRANSPLANTATION (SCT) (HR patients with matched family [MFD] or unrelated donor):

CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily on days -5 to -2.

TRANSPLANTATION: Patients undergo allogeneic SCT within 36 to 48 hours after the last dose of busulfan.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or PO beginning on day -2 and continuing until day 98 (matched sibling donor) or day 180 (with taper) (other related/unrelated donors or cord blood) and methotrexate IV on days 1, 3, and 6 (matched sibling/cord blood donors) or days 1, 3, 6, and 11 (other related/unrelated donors). Patients with unrelated donors also receive antithymocyte globulin IV over 6-8 hours on days -3 to -1.

MAINTENANCE: Patients receive sorafenib tosylate PO starting on day 40-100 after completion of intensification II or SCT for one year.

ARM C (COHORT 2):

INDUCTION I: Patients receive cytarabine IT and ADE chemotherapy as in Arm A, Induction I and sorafenib tosylate PO at the time of known HR FLT3/ITD+ (including in Induction I and concurrently with chemotherapy).

INDUCTION II: Patients receive cytarabine IT on day 1, cytarabine IV over 1-30 minutes on days 1-8, daunorubicin hydrochloride IV over 1-15 minutes on days 1, 3, and 5, etoposide IV over 1-2 hours on days 1-5, and sorafenib tosylate PO on days 9-36.

INTENSIFICATION I: Patients receive cytarabine IT and AE chemotherapy in Arm A, Intensification II, and sorafenib tosylate PO on daily on days 6-28.

INTENSIFICATION II: Patients receive cytarabine IT on day 1, MA chemotherapy as in Arm A, Induction II (HR patients), and sorafenib tosylate PO on days 7-34.

STEM CELL TRANSPLANTATION (SCT) (HR patients with matched family [MFD] or unrelated donor):

CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily on days -5 to -2.

TRANSPLANTATION: Patients undergo allogeneic SCT within 36 to 48 hours after the last dose of busulfan.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or PO beginning on day -2 and continuing until day 98 (matched sibling donor) or day 180 (with taper) (other related/unrelated donors or cord blood) and methotrexate IV on days 1, 3, and 6 (matched sibling/cord blood donors) or days 1, 3, 6, and 11 (other related/unrelated donors). Patients with unrelated donors also receive antithymocyte globulin IV over 6-8 hours on days -3 to -1.

MAINTENANCE: Patients receive sorafenib tosylate PO starting on day 40-100 after completion of intensification II or SCT for one year.

ARM C (COHORT 3):

INDUCTION I: Patients receive cytarabine IT and ADE chemotherapy as in Arm A, Induction I and sorafenib tosylate PO on days 11-28.

INDUCTION II: Patients receive cytarabine IT on day 1, cytarabine IV over 1-30 minutes on days 1-8, daunorubicin hydrochloride IV over 1-15 minutes on days 1, 3, and 5, etoposide IV over 1-2 hours on days 1-5, and sorafenib tosylate PO on days 9-36.

INTENSIFICATION I: Patients receive cytarabine IT and AE chemotherapy in Arm A, Intensification II, and sorafenib tosylate PO on daily on days 6-28.

INTENSIFICATION II: Patients receive cytarabine IT on day 1, MA chemotherapy as in Arm A, Induction II (HR patients), and sorafenib tosylate PO on days 7-34.

STEM CELL TRANSPLANTATION (SCT) (HR patients with matched family [MFD] or unrelated donor):

CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily on days -5 to -2.

TRANSPLANTATION: Patients undergo allogeneic SCT within 36 to 48 hours after the last dose of busulfan.

GVHD PROPHYLAXIS: Patients receive tacrolimus IV continuously or PO beginning on day -2 and continuing until day 98 (matched sibling donor) or day 180 (with taper) (other related/unrelated donors or cord blood) and methotrexate IV on days 1, 3, and 6 (matched sibling/cord blood donors) or days 1, 3, 6, and 11 (other related/unrelated donors). Patients with unrelated donors also receive antithymocyte globulin IV over 6-8 hours on days -3 to -1.

MAINTENANCE: Patients receive sorafenib tosylate PO starting on day 40-100 after completion of intensification II or SCT for one year.

ARM D:

INDUCTION I: Patients with unknown FLT3/ITD status prior to study enrollment receive cytarabine IT and ADE chemotherapy as in Arm A, Induction I. If patients are determined to be HR FLT3/ITD+ no later than the end of Induction I they will be eligible to participate in Arm C.

After completion of study therapy, patients are followed up monthly for 6 months, every 2 months for 6 months, every 4 months for 1 year, every 6 months for 1 year, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with de novo acute myelogenous leukemia
* Patients with previously untreated primary AML who meet the customary criteria for AML with >= 20% bone marrow blasts as set out in the 2008 World Health Organization (WHO) Myeloid Neoplasm Classification are eligible

  * Attempts to obtain bone marrow either by aspirate or biopsy must be made unless clinically prohibitive; in cases where it is clinically prohibitive, peripheral blood with an excess of 20% blasts and in which adequate flow cytometric and cytogenetics/fluorescent in situ hybridization (FISH) testing is feasible can be substituted for the marrow exam at diagnosis
* Patients with < 20% bone marrow blasts are eligible if they have:

  * A karyotypic abnormality characteristic of de novo AML (t(8;21)(q22;q22), inv(16)(p13q22) or t(16;16)(p13;q22) or 11q23 abnormalities
  * The unequivocal presence of megakaryoblasts, or
  * Biopsy proven isolated myeloid sarcoma (myeloblastoma; chloroma, including leukemia cutis)
* Patients with any performance status are eligible for enrollment
* Prior therapy with hydroxyurea, all-trans retinoic acid (ATRA), corticosteroids (any route), and IT cytarabine given at diagnosis is allowed; hydroxyurea and ATRA must be discontinued prior to initiation of protocol therapy; patients who have previously received any other chemotherapy, radiation therapy or any other antileukemic therapy are not eligible for this protocol

Exclusion Criteria:

* Patients with any of the following constitutional conditions are not eligible:

  * Fanconi anemia
  * Shwachman syndrome
  * Any other known bone marrow failure syndrome
  * Patients with constitutional trisomy 21 or with constitutional mosaicism of trisomy 21 Note: enrollment may occur pending results of clinically indicated studies to exclude these conditions
* Patients with any of the following oncologic diagnoses are not eligible:

  * Any concurrent malignancy
  * Juvenile myelomonocytic leukemia (JMML)
  * Philadelphia chromosome positive AML
  * Biphenotypic or bilineal acute leukemia
  * Acute promyelocytic leukemia
  * Acute myeloid leukemia arising from myelodysplasia
  * Therapy-related myeloid neoplasms Note: enrollment may occur pending results of clinically indicated studies to exclude these conditions
* Pregnancy and breast feeding
* Female patients who are pregnant are ineligible
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1645 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2027-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Aplenc, Principal Investigator — Children's Oncology Group
Locations (220):
- United States (195):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Huang BJ, Meyer LK, Alonzo TA, Wang YC, Lamble AJ, Ries RE, Wang W, Hirsch B, Raca G, Ma X, Gamis AS, Aplenc R, Kolb EA, Cooper TM, Tarlock K, Loken MR, Meshinchi S, Chewning JH, Woods WG, Horan JT. Hematopoietic Stem Cell Transplantation Outcomes for High-Risk AML: A Report From the Children's Oncology Group. J Clin Oncol. 2025 Jun 10;43(17):1961-1971. doi: 10.1200/JCO-24-01841. Epub 2025 Apr 28. PMID 40294366
- [Derived] Tarlock K, Gerbing RB, Ries RE, Smith JL, Leonti A, Huang BJ, Kirkey D, Robinson L, Peplinski JH, Lange B, Cooper TM, Gamis AS, Kolb EA, Aplenc R, Pollard JA, Alonzo TA, Meshinchi S. Prognostic impact of cooccurring mutations in FLT3-ITD pediatric acute myeloid leukemia. Blood Adv. 2024 May 14;8(9):2094-2103. doi: 10.1182/bloodadvances.2023011980. PMID 38295280
- [Derived] Zarnegar-Lumley S, Alonzo TA, Gerbing RB, Othus M, Sun Z, Ries RE, Wang J, Leonti A, Kutny MA, Ostronoff F, Radich JP, Appelbaum FR, Pogosova-Agadjanyan EL, O'Dwyer K, Tallman MS, Litzow M, Atallah E, Cooper TM, Aplenc RA, Abdel-Wahab O, Gamis AS, Luger S, Erba H, Levine R, Kolb EA, Stirewalt DL, Meshinchi S, Tarlock K. Characteristics and prognostic impact of IDH mutations in AML: a COG, SWOG, and ECOG analysis. Blood Adv. 2023 Oct 10;7(19):5941-5953. doi: 10.1182/bloodadvances.2022008282. PMID 37267439
- [Derived] Bertrums EJM, Smith JL, Harmon L, Ries RE, Wang YJ, Alonzo TA, Menssen AJ, Chisholm KM, Leonti AR, Tarlock K, Ostronoff F, Pogosova-Agadjanyan EL, Kaspers GJL, Hasle H, Dworzak M, Walter C, Muhlegger N, Morerio C, Pardo L, Hirsch B, Raimondi S, Cooper TM, Aplenc R, Gamis AS, Kolb EA, Farrar JE, Stirewalt D, Ma X, Shaw TI, Furlan SN, Brodersen LE, Loken MR, Van den Heuvel-Eibrink MM, Zwaan CM, Triche TJ, Goemans BF, Meshinchi S. Comprehensive molecular and clinical characterization of NUP98 fusions in pediatric acute myeloid leukemia. Haematologica. 2023 Aug 1;108(8):2044-2058. doi: 10.3324/haematol.2022.281653. PMID 36815378
- [Derived] Pollard JA, Alonzo TA, Gerbing R, Brown P, Fox E, Choi J, Fisher B, Hirsch B, Kahwash S, Getz K, Levine J, Brodersen LE, Loken MR, Raimondi S, Tarlock K, Wood A, Sung L, Kolb EA, Gamis A, Meshinchi S, Aplenc R. Sorafenib in Combination With Standard Chemotherapy for Children With High Allelic Ratio FLT3/ITD+ Acute Myeloid Leukemia: A Report From the Children's Oncology Group Protocol AAML1031. J Clin Oncol. 2022 Jun 20;40(18):2023-2035. doi: 10.1200/JCO.21.01612. Epub 2022 Mar 29. PMID 35349331
- [Derived] Lamble AJ, Eidenschink Brodersen L, Alonzo TA, Wang J, Pardo L, Sung L, Cooper TM, Kolb EA, Aplenc R, Tasian SK, Loken MR, Meshinchi S. CD123 Expression Is Associated With High-Risk Disease Characteristics in Childhood Acute Myeloid Leukemia: A Report From the Children's Oncology Group. J Clin Oncol. 2022 Jan 20;40(3):252-261. doi: 10.1200/JCO.21.01595. Epub 2021 Dec 2. PMID 34855461
- [Derived] Elgarten CW, Wood AC, Li Y, Alonzo TA, Brodersen LE, Gerbing RB, Getz KD, Huang YV, Loken M, Meshinchi S, Pollard JA, Sung L, Woods WG, Kolb EA, Gamis AS, Aplenc R. Outcomes of intensification of induction chemotherapy for children with high-risk acute myeloid leukemia: A report from the Children's Oncology Group. Pediatr Blood Cancer. 2021 Dec;68(12):e29281. doi: 10.1002/pbc.29281. Epub 2021 Oct 1. PMID 34596937
- [Derived] Aplenc R, Meshinchi S, Sung L, Alonzo T, Choi J, Fisher B, Gerbing R, Hirsch B, Horton T, Kahwash S, Levine J, Loken M, Brodersen L, Pollard J, Raimondi S, Kolb EA, Gamis A. Bortezomib with standard chemotherapy for children with acute myeloid leukemia does not improve treatment outcomes: a report from the Children's Oncology Group. Haematologica. 2020 Jul;105(7):1879-1886. doi: 10.3324/haematol.2019.220962. Epub 2020 Feb 6. PMID 32029509
- [Derived] Garcia-Pavia P, Kim Y, Restrepo-Cordoba MA, Lunde IG, Wakimoto H, Smith AM, Toepfer CN, Getz K, Gorham J, Patel P, Ito K, Willcox JA, Arany Z, Li J, Owens AT, Govind R, Nunez B, Mazaika E, Bayes-Genis A, Walsh R, Finkelman B, Lupon J, Whiffin N, Serrano I, Midwinter W, Wilk A, Bardaji A, Ingold N, Buchan R, Tayal U, Pascual-Figal DA, de Marvao A, Ahmad M, Garcia-Pinilla JM, Pantazis A, Dominguez F, John Baksi A, O'Regan DP, Rosen SD, Prasad SK, Lara-Pezzi E, Provencio M, Lyon AR, Alonso-Pulpon L, Cook SA, DePalma SR, Barton PJR, Aplenc R, Seidman JG, Ky B, Ware JS, Seidman CE. Genetic Variants Associated With Cancer Therapy-Induced Cardiomyopathy. Circulation. 2019 Jul 2;140(1):31-41. doi: 10.1161/CIRCULATIONAHA.118.037934. Epub 2019 Apr 16. PMID 30987448
- [Derived] Lin KH, Xie A, Rutter JC, Ahn YR, Lloyd-Cowden JM, Nichols AG, Soderquist RS, Koves TR, Muoio DM, MacIver NJ, Lamba JK, Pardee TS, McCall CM, Rizzieri DA, Wood KC. Systematic Dissection of the Metabolic-Apoptotic Interface in AML Reveals Heme Biosynthesis to Be a Regulator of Drug Sensitivity. Cell Metab. 2019 May 7;29(5):1217-1231.e7. doi: 10.1016/j.cmet.2019.01.011. Epub 2019 Feb 14. PMID 30773463
- [Derived] Hanley MJ, Mould DR, Taylor TJ, Gupta N, Suryanarayan K, Neuwirth R, Esseltine DL, Horton TM, Aplenc R, Alonzo TA, Lu X, Milton A, Venkatakrishnan K. Population Pharmacokinetic Analysis of Bortezomib in Pediatric Leukemia Patients: Model-Based Support for Body Surface Area-Based Dosing Over the 2- to 16-Year Age Range. J Clin Pharmacol. 2017 Sep;57(9):1183-1193. doi: 10.1002/jcph.906. Epub 2017 Apr 18. PMID 28419486
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results in the Participant Flow table summarize final (or analysis) arm assignment. Therefore, results for patients on Arms A, B, and D do not include any patient who transferred to Arm C.
Groups:
- Arm A: INDUCTION (IND) 1Pts receive intrathecal (IT) cytarabine on day 1 and ADE with IV cytarabine over 1-30 minutes on days 1-10; daunorubicin hydrochloride IV over 1-15 minutes days1, 3, 5; etoposide IV 1-2 hours days 1-5.
  IND IILow risk (LR) pts receive cytarabine IT and ADE chemotherapy as in INDI. High risk (HR) cytarabine IT day 1, MA chemo comprising high-dose cytarabine IV over 1-3 hours days1-4, mitoxantrone IV over 15-30 minutes days 3-6. INTENSIFICATION (INT) I: cytarabine IT day 1, AE chemo with high-dose cytarabine IV over 1-3 hours, etoposide IV over 1-2 hours days 1-5. INT II: LR-cytarabine IT day 1; Induction II MA chemo. HR and no SCT donor - high-dose cytarabine IV over 3 hours days1, 2, 8, 9; asparaginase intramuscularly (IM) days 2,9.
  SCT:
  pts receive fludarabine phosphate IV over 30 minutes once daily days -5 to -2, busulfan IV over 2 hours 4 times daily days -5 to -2.
  Allogeneic SCT within 36 to 48 hours after last busulfan dose. Pts receive GVHD prophylaxis.
- Arm B: IND I: Pts receive cytarabine IT and ADE chemotherapy as in Induction I, Arm A. Patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8.
  IND II: LR pts receive cytarabine IT, ADE chemotherapy, bortezomib as in IND I. HR pts receive cytarabine IT, MA as in IND II, Arm A (HR patients) and bortezomib IV on days 1, 4, 8.
  INT I: Pts receive cytarabine IT and AE in Arm A, Intensification II, and bortezomib IV on days 1, 4, 8. INT II: LR pts receive cytarabine IT on day 1, MA as in Arm A, IND II (HR patients), and bortezomib IV on days 1, 4, 8. HR pts with no donor for SCT receive high-dose cytarabine IV over 3 hours on days 1, 2, 8, 9 and asparaginase intramuscularly (IM) on days 2 and 9.
  SCT - Pts receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily on days -5 to -2.Pts undergo allogeneic SCT within 36 to 48 hours after the last dose of busulfan. Pts receive GVHD prophylaxis.
- Arm C (Cohort 1): IND II: Pts receive cytarabine IT on day 1, cytarabine IV over 1-30 minutes on days 1-8, daunorubicin hydrochloride IV over 1-15 minutes on days 1, 3, and 5, etoposide IV over 1-2 hours on days 1-5, sorafenib tosylate PO on days 9-36.
  INT I: Pts receive cytarabine IT and AE chemotherapy in Arm A, Intensification II, and sorafenib tosylate PO on daily on days 6-28.
  INT II: Pts receive cytarabine IT on day 1, MA chemotherapy as in Arm A, Induction II (HR patients), sorafenib tosylate PO on days 7-34.
  SCT (HR patients with matched family [MFD] or unrelated donor):
  Pts receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2, busulfan IV over 2 hours 4 times daily on days -5 to -2.
  Patients undergo allogeneic SCT within 36 to 48 hours after the last dose of busulfan. Pts receive GVHD prophylaxis.
  MAINTENANCE: Pts receive sorafenib tosylate PO starting day 40-100 after INT II or SCT for one year.
- Arm C (Cohort 2): IND I: Pts receive cytarabine IT & ADE as in Arm A, IND I & sorafenib tosylate PO at the time of known HR FLT3/ITD+ (including IND I & concurrently with chemo).
  IND II: Pts receive cytarabine IT day (d) 1, cytarabine IV over 1-30 minutes on d 1-8, daunorubicin hydrochloride IV over 1-15 minutes days 1, 3, 5, etoposide IV over 1-2 hours d 1-5, sorafenib tosylate PO d 9-36.
  INT I: Pts receive cytarabine IT and AE as in Arm A, INT II, and sorafenib tosylate PO on daily d 6-28.
  INT II: Pts receive cytarabine IT on d 1, MA as in Arm A, IND II (HR pts), sorafenib tosylate PO d 7-34.
  SCT (HR patients with matched family [MFD] or unrelated donor):
  Pts receive fludarabine phosphate IV over 30 minutes once daily on d -5 to -2, busulfan IV over 2 hours 4 times daily d -5 to -2.
  Pts undergo allogeneic SCT within 36-48 hours after last busulfan dose. Pts receive GVHD prophylaxis. MAINTENANCE: Pts receive sorafenib tosylate PO starting d 40-100 after INT II or SCT for 1 year.
- Arm C (Cohort 3): IND I: Pts receive cytarabine IT & ADE as in Arm A, IND I & sorafenib tosylate PO days 11-28.
  IND II: Pts receive cytarabine IT day 1, cytarabine IV over 1-30 minutes on days 1-8, daunorubicin hydrochloride IV over 1-15 minutes days 1, 3, 5, etoposide IV over 1-2 hours days 1-5, sorafenib tosylate PO days 9-36.
  INT I: Pts receive cytarabine IT & AE as in Arm A, INT II, & sorafenib tosylate PO daily days 6-28.
  INT II: Pts receive cytarabine IT day 1, MA as in Arm A, IND II (HR patients), & sorafenib tosylate PO days 7-34.
  SCT (HR patients with matched family [MFD] or unrelated donor):
  Pts receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily days -5 to -2.
  Pts undergo allogeneic SCT within 36 to 48 hours after last busulfan dose. Pts receive GVHD prophylaxis. MAINTENANCE: Pts receive sorafenib tosylate PO starting day 40-100 after INT II or SCT for 1 year.
- Arm D: INDUCTION I: Patients with unknown FLT3/ITD status prior to study enrollment receive cytarabine IT and ADE chemotherapy as in Arm A, Induction I. If patients are determined to be HR FLT3/ITD+ no later than the end of Induction I they will be eligible to participate in Arm C.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2) | Arm C (Cohort 3) | Arm D
Started | 580 | 591 | 12 | 33 | 47 | 382
Completed | 396 | 399 | 6 | 12 | 15 | 368
Not Completed | 184 | 192 | 6 | 21 | 32 | 14
Not completed — Adverse Event | 12 | 17 | 0 | 4 | 1 | 0
Not completed — Death | 22 | 16 | 0 | 0 | 2 | 2
Not completed — Lack of Efficacy | 69 | 61 | 4 | 8 | 5 | 0
Not completed — Physician Decision | 48 | 63 | 1 | 7 | 14 | 3
Not completed — Withdrawal by Subject | 12 | 19 | 1 | 2 | 10 | 3
Not completed — Ineligible | 19 | 13 | 0 | 0 | 0 | 4
Not completed — Did not start treatment | 2 | 3 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm A: INDUCTION (IND) 1Pts receive intrathecal (IT) cytarabine on day 1 and ADE with IV cytarabine over 1-30 minutes on days 1-10; daunorubicin hydrochloride IV over 1-15 minutes days1, 3, 5; etoposide IV 1-2 hours days1-5.
  IND IILow risk (LR) pts receive cytarabine IT and ADE chemotherapy as in INDI. High risk (HR) cytarabine IT day 1, MA chemo comprising high-dose cytarabine IV over 1-3 hours days1-4, mitoxantrone IV over 15-30 minutes days 3-6. INTENSIFICATION (INT) I: cytarabine IT day 1, AE chemo with high-dose cytarabine IV over 1-3 hours, etoposide IV over 1-2 hours days 1-5. INT II: LR-cytarabine IT day 1; Induction II MA chemo. HR and no SCT donor - high-dose cytarabine IV over 3 hours days1, 2, 8, 9; asparaginase intramuscularly (IM) days2,9.
  SCT:
  : pts receive fludarabine phosphate IV over 30 minutes once daily days -5 to -2, busulfan IV over 2 hours 4 times daily days -5 to -2.
  Allogeneic SCT within 36 to 48 hours after last busulfan dose. Pts receive GVHD prophylaxis.
- Arm C (Cohort 2): IND I: Pts receive cytarabine IT & ADE as in Arm A, IND I & sorafenib tosylate PO at the time of known HR FLT3/ITD+ (including IND I & concurrently with chemo).
  IND II: Pts receive cytarabine IT day (d) 1, cytarabine IV over 1-30 minutes on d 1-8, daunorubicin hydrochloride IV over 1-15 minutes days 1, 3, 5, etoposide IV over 1-2 hours d 1-5, sorafenib tosylate PO d 9-36.
  INTE I: Pts receive cytarabine IT and AE in Arm A, INT II, and sorafenib tosylate PO on daily d 6-28.
  INT II: Pts receive cytarabine IT on d 1, MA as in Arm A, IND II (HR pts), sorafenib tosylate PO d 7-34.
  SCT (HR patients with matched family [MFD] or unrelated donor):
  Pts receive fludarabine phosphate IV over 30 minutes once daily on d -5 to -2, busulfan IV over 2 hours 4 times daily d -5 to -2.
  Pts undergo allogeneic SCT within 36-48 hours after last busulfan dose. Pts receive GVHD prophylaxis. MAINTENANCE: Pts receive sorafenib tosylate PO starting d 40-100 after INT II or SCT for 1 year.
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2) | Arm C (Cohort 3) | Arm D | Total
Number analyzed (Participants) | 580 | 591 | 12 | 33 | 47 | 382 | 1645
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5940 (6.6172) | 9.4322 (6.6408) | 11.7930 (4.9715) | 12.4961 (5.0103) | 11.7907 (5.0134) | 9.1600 (6.6186) | 9.5721 (6.5691)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 305 | 8 | 18 | 20 | 203 | 858
  Male | 276 | 286 | 4 | 15 | 27 | 179 | 787
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 107 | 106 | 1 | 5 | 3 | 80 | 302
  Not Hispanic or Latino | 457 | 465 | 10 | 28 | 36 | 273 | 1269
  Unknown or Not Reported | 16 | 20 | 1 | 0 | 8 | 29 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 0 | 0 | 1 | 2 | 12
  Asian | 27 | 28 | 0 | 2 | 1 | 21 | 79
  Native Hawaiian or Other Pacific Islander | 3 | 6 | 0 | 0 | 0 | 4 | 13
  Black or African American | 76 | 70 | 4 | 3 | 5 | 40 | 198
  White | 411 | 413 | 7 | 27 | 33 | 257 | 1148
  More than one race | 0 | 1 | 0 | 0 | 1 | 6 | 8
  Unknown or Not Reported | 60 | 67 | 1 | 1 | 6 | 52 | 187
Region of Enrollment [Number; unit: participants]
  United States | 514 | 515 | 11 | 29 | 41 | 334 | 1444
  Canada | 31 | 43 | 1 | 3 | 5 | 24 | 107
  Australia | 23 | 29 | 0 | 1 | 1 | 15 | 69
  New Zealand | 12 | 4 | 0 | 0 | 0 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) for Patients Without High Allelic Ratio FLT3/ITD+ Mutations
Description: The Kaplan-Meier method will be used to estimate 3-year EFS, defined as the time from study entry until induction failure, relapse, secondary malignancy, or death.
Time Frame: Up to 3 years
Population: Patients ineligible, did not start treatment, or on Arm D are excluded from analyses of EFS. Arm D patients who were not eligible for Arm C by the end of induction I were declared off study per protocol; thus, no outcome data were collected for Arm D patients. Arms A and B are limited to patients without high allelic ratio FLT3/ITD+ mutations.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 540 | 552
percentage of patients | 45.64 [41.34 to 49.83] | 46.95 [42.69 to 51.09]

2. Primary Outcome: EFS for Patients on Arm C, Cohort 1
Description: as for outcome 1
Time Frame: Up to 3 years
Population: Patients ineligible, did not start treatment, or on Arm D are excluded from analyses of EFS. Arm D patients who were not eligible for Arm C by the end of induction I were declared off study per protocol; thus, no outcome data were collected for Arm D patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm C (Cohort 1)
Number analyzed (Participants) | 12
percentage of patients | 25.00 [6.01 to 50.48]

3. Primary Outcome: EFS for Patients on Arm C, Cohort 2
Description: as for outcome 1
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm C (Cohort 2)
Number analyzed (Participants) | 33
percentage of patients | 56.12 [37.33 to 71.28]

4. Primary Outcome: EFS for Patients on Arm C, Cohort 3
Description: as for outcome 1
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm C (Cohort 3)
Number analyzed (Participants) | 47
percentage of patients | 58.18 [42.30 to 71.11]

5. Secondary Outcome: Overall Survival (OS) for Patients Without High Allelic Ratio FLT3/ITD+ Mutations
Description: The Kaplan-Meier method will be used to estimate 3-year OS, defined as the time from study entry until death.
Time Frame: Up to 3 years
Population: Patients ineligible, did not start treatment, or on Arm D are excluded from analyses of OS. Arm D patients who were not eligible for Arm C by the end of induction I were declared off study per protocol; thus, no outcome data were collected for Arm D patients. Arms A and B are limited to patients without high allelic ratio FLT3/ITD+ mutations.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 540 | 552
percentage of patients | 65.04 [60.75 to 68.98] | 68.45 [64.33 to 72.21]

6. Secondary Outcome: OS for Patients on Arm C, Cohort 1
Description: The Kaplan-Meier method will be used to estimate 3-year OS, defined as the time from study entry until death.
Time Frame: Up to 3 years
Population: Patients ineligible, did not start treatment, or on Arm D are excluded from analyses of OS. Arm D patients who were not eligible for Arm C by the end of induction I were declared off study per protocol; thus, no outcome data were collected for Arm D patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm C (Cohort 1)
Number analyzed (Participants) | 12
percentage of patients | 41.67 [15.25 to 66.53]

7. Secondary Outcome: OS for Patients on Arm C, Cohort 2
Description: The Kaplan-Meier method will be used to estimate 3-year OS, defined as the time from study entry until death.
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm C (Cohort 2)
Number analyzed (Participants) | 33
percentage of patients | 64.77 [45.37 to 78.77]

8. Secondary Outcome: OS for Patients on Arm C, Cohort 3
Description: The Kaplan-Meier method will be used to estimate 3-year OS, defined as the time from study entry until death.
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm C (Cohort 3)
Number analyzed (Participants) | 47
percentage of patients | 61.84 [44.09 to 75.42]

9. Secondary Outcome: Relapse Rate for Patients Without High Allelic Ratio FLT3/ITD+ Mutations
Description: Cumulative incidence estimates 3 year relapse rate defined as time from study entry to induction failure or relapse where deaths or secondary malignancies are competing events.
Time Frame: Up to 3 years
Population: Patients ineligible, did not start treatment, or on Arms C or D are excluded. Arm D patients who were not eligible for Arm C by the end of induction I were declared off study per protocol; thus, no outcome data were collected for Arm D patients. Results are limited to patients on Arms A and B without high allelic ratio FLT3/ITD+ mutations.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 540 | 552
percentage of patients | 46.67 [42.36 to 50.86] | 46.65 [42.39 to 50.80]

10. Secondary Outcome: Proportion of Patients Experiencing Grade 3 or Higher Non-hematologic Toxicities and Infections While on Protocol Therapy
Description: The proportion of patients experiencing at least one grade 3 or higher non-hematologic toxicity and infection while on protocol therapy will be estimated along with the corresponding 95% confidence interval determined using a binomial exact method. Toxicity will be assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).
Time Frame: Up to 2 years
Population: Patients ineligible or who did not start treatment are excluded from results.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2) | Arm C (Cohort 3) | Arm D
Number analyzed (Participants) | 559 | 575 | 12 | 33 | 47 | 376
Proportion of patients | 0.8819 [0.8522 to 0.9075] | 0.9217 [0.8967 to 0.9423] | 0.9167 [0.6152 to 0.9979] | 0.9394 [0.7977 to 0.9926] | 0.9149 [0.7962 to 0.9763] | 0.0239 [0.0110 to 0.0450]

11. Secondary Outcome: Proportion of High Risk Children Without HR FLT3/ITD+ Converting From Positive MRD at End of Induction I to Negative MRD at the End of Induction II
Description: The proportion of high risk children without HR FLT3/ITD+ converting from positive MRD at end of Induction I to negative MRD at the end of Induction II will be estimated as well as the corresponding 95% confidence interval determined using a binomial exact method.
Time Frame: Up to 8 weeks
Population: Patients ineligible, did not start treatment, on Arms C, D are excluded from results. Complete MRD results were not collected for Arm D patients due to being declared off study at end of induction I. Results limited to High Risk patients without high allelic ratio FLT3/ITD+ mutations and with evaluable MRD data from end of Induction I and II.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 76 | 84
Proportion of patients | 0.5000 [0.3830 to 0.6170] | 0.5238 [0.4119 to 0.6340]

12. Secondary Outcome: Total Scale Score From Parent-reported Pediatric Quality of Life Inventory Module
Description: Results represent the total scale scores from the parent report of the PedsQL™ 4.0 Generic Core Scales for timepoint 1 (up to 14 days from start of therapy). Items are reverse-scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Therefore, a higher number is a better outcome. The total score is the sum of all the items divided by the number of items answered on all the scales. "Scores on a scale" is used for a unit of measure.
Time Frame: Up to 14 days
Population: Patients ineligible or who did not start treatment are excluded from results. Patients on Arms C (cohort 3) or Arm D are excluded due to enrolling post quality of life study accrual completion. Results are limited to only patients with an evaluable total scale score.
Measure: Mean (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2)
Number analyzed (Participants) | 228 | 195 | 8 | 16
Scores on a scale | 68.3 [55.7 to 81.5] | 67.8 [52.2 to 83.7] | 71.3 [58.7 to 87.5] | 61.6 [46.2 to 81.0]

13. Secondary Outcome: Total Scale Score From Parent-reported Cancer Module
Description: Results represent the total scale scores from the parent report of the PedsQL™ 3.0 Cancer Module for timepoint 1 (up to 14 days from start of therapy). Items are reverse-scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Therefore, a higher number is a better outcome. The total score is the sum of all the items divided by the number of items answered on all the scales. "Scores on a scale" is used for a unit of measure.
Time Frame: Up to 14 days
Population: as for outcome 12
Measure: Mean (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2)
Number analyzed (Participants) | 230 | 193 | 8 | 16
Scores on a scale | 66.2 [53.7 to 78.7] | 65.8 [53.7 to 77.9] | 74.9 [69.0 to 81.7] | 63.7 [56.9 to 74.0]

14. Secondary Outcome: Total Scale Score From Parent-reported Multidimensional Fatigue Scale Module
Description: Results represent the total scale scores from the parent report of the PedsQL™ Multidimensional Fatigue Scale for timepoint 1 (up to 14 days from start of therapy). Items are reverse-scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Therefore, a higher number is a better outcome. The total score is the sum of all the items divided by the number of items answered on all the scales. "Scores on a scale" is used for a unit of measure.
Time Frame: Up to 14 days
Population: as for outcome 12
Measure: Mean (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2)
Number analyzed (Participants) | 226 | 194 | 8 | 16
Scores on a scale | 60.5 [45.8 to 75.0] | 58.1 [44.4 to 73.6] | 71.2 [52.8 to 87.5] | 48.2 [30.6 to 64.6]

15. Secondary Outcome: Bortezomib Clearance
Description: Median and range of bortezomib clearance during Induction II.
Time Frame: Day 8 of Induction II
Population: Only eligible patients on Arm B with evaluable Bortezomib PK clearance data during Induction II are reported.
Measure: Median (Full Range); unit: Liters/hour/m^2
Arm/Group | Arm B
Number analyzed (Participants) | 53
Liters/hour/m^2 | 8.42 [3.52 to 12.70]

16. Secondary Outcome: Sorafenib Steady State Concentration
Description: Median and range of sorafenib steady state concentration for Induction I.
Time Frame: Up to 30 days
Population: Data reported from Arm C were collected and analyzed regardless of the cohort as pre-specified in the study protocol. Only eligible patients on Arm C with evaluable Sorafenib steady state concentration data during Induction I are reported.
Measure: Median (Full Range); unit: Nanogram/Milliliter
Groups:
- Arm C: Arm C (Cohort 1) IND II:cytarabine IT; cytarabine IV; daunorubicin hydrochloride IV; etoposide IV; sorafenib tosylate PO INT I:cytarabine IT; AE chemotherapy as Arm A, Intensification II; sorafenib tosylate PO INT II:cytarabine IT; MA chemotherapy as Arm A, Induction II (HR patients); sorafenib tosylate PO.
  SCT (HR pts w/ matched family [MFD] or unrelated donor): fludarabine phosphate IV; busulfan IV; allogeneic SCT; GVHD prophylaxis.
  MAINTENANCE:sorafenib tosylate PO
  Arm C (Cohort 2 and 3) IND I:cytarabine IT; ADE as Arm A, IND I; sorafenib tosylate PO IND II:cytarabine IT; cytarabine IV; daunorubicin hydrochloride IV; etoposide IV; sorafenib tosylate PO INT I:cytarabine IT; AE as Arm A, INT II, & sorafenib tosylate PO INT II:cytarabine IT; MA as Arm A, IND II (HR patients); sorafenib tosylate PO. SCT (HR pts w/ matched family [MFD] or unrelated donor): fludarabine phosphate IV; busulfan IV; allogeneic SCT; GVHD prophylaxis.
  MAINTENANCE:sorafenib tosylate PO
Arm/Group | Arm C
Number analyzed (Participants) | 23
Nanogram/Milliliter | 1090.0 [290.0 to 4740.0]

17. Secondary Outcome: Change in Shortening Fraction
Description: Mean percentage change in shortening fraction from baseline to the end of Induction I will be determined for eligible patients enrolled on Arms A, B and C.
Time Frame: Up to 4 weeks
Population: Patients ineligible, did not start treatment, or on Arm D are excluded from results. Shortening fraction data were not collected at end of Induction I for patients enrolled to Arm D. Results are limited to patients with evaluable shortening fraction data from study entry and at end of Induction I .
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2) | Arm C (Cohort 3)
Number analyzed (Participants) | 499 | 503 | 9 | 32 | 41
Percentage change | -1.8445 (5.2070) | -2.6298 (6.7797) | -2.2333 (4.7689) | -3.6700 (5.3115) | -3.4246 (4.8583)

18. Secondary Outcome: Change in Ejection Fraction
Description: The mean percentage change in ejection fraction from baseline to the end of Induction I will be determined for eligible patients enrolled on Arms A, B and C.
Time Frame: Up to 4 weeks
Population: Patients ineligible, did not start treatment, or on Arm D are excluded from results. Ejection fraction data were not collected at end of Induction I for patients enrolled to Arm D. Results are limited to patients with evaluable ejection fraction data from study entry and at end of Induction I .
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2) | Arm C (Cohort 3)
Number analyzed (Participants) | 426 | 425 | 6 | 30 | 38
Percentage change | -2.0272 (7.1843) | -2.3453 (7.6974) | -7.5000 (12.5340) | -5.1997 (7.0532) | -3.4624 (6.7516)

19. Secondary Outcome: Serum Concentrations of GVHD Biomarker
Description: The mean serum concentration of the day 28 GVHD biomarker will be estimated as well as the corresponding 95% confidence interval.
Time Frame: Up to day 28 after SCT
Population: Data were never collected
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2) | Arm C (Cohort 3)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Other Pre Specified Outcome: Course Duration
Description: Descriptive statistics will be used to summarize length of hospitalization time.
Time Frame: Up to 6 months
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Incidence of Treatment-related Mortality
Description: Cumulative incidence estimates that account for competing events will be used to estimate treatment-related mortality.
Time Frame: Up to 2 years
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Length of Hospitalization
Description: Descriptive statistics will be used to summarize length of hospitalization time.
Time Frame: Up to 6 months
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Remission Rate After 1 Course of Therapy
Description: The proportion of patients achieving remission after 1 course of therapy will be estimated along with a corresponding 95% confidence interval.
Time Frame: 4 weeks
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Remission Rate After 2 Courses of Therapy
Description: The proportion of patients achieving remission after 2 courses of therapy will be estimated along with a corresponding 95% confidence interval.
Time Frame: 8 weeks
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Time to Blood Count Recovery
Description: Cumulative incidence estimates that account for competing events will be used to estimate time to count recovery.
Time Frame: Up to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: While patients were on protocol therapy (including up to 4 courses, stem cell transplant course, and 3 courses of maintenance therapy)) or up to 7 years in follow-up.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Groups:
- Arm C (Cohort 3): IND I: Pts receive cytarabine IT & ADE as in Arm A, IND I & sorafenib tosylate PO days 11-28.
  IND II: Pts receive cytarabine IT day 1, cytarabine IV over 1-30 minutes on days 1-8, daunorubicin hydrochloride IV over 1-15 minutes days 1, 3, 5, etoposide IV over 1-2 hours days 1-5, sorafenib tosylate PO days 9-36.
  INT I: Pts receive cytarabine IT & AE cin Arm A, INT II, & sorafenib tosylate PO daily days 6-28.
  INT II: Pts receive cytarabine IT day 1, MA as in Arm A, IND II (HR patients), & sorafenib tosylate PO days 7-34.
  SCT (HR patients with matched family [MFD] or unrelated donor):
  Pts receive fludarabine phosphate IV over 30 minutes once daily on days -5 to -2 and busulfan IV over 2 hours 4 times daily days -5 to -2.
  Pts undergo allogeneic SCT within 36 to 48 hours after last busulfan dose. Pts receive GVHD prophylaxis. MAINTENANCE: Pts receive sorafenib tosylate PO starting day 40-100 after INT II or SCT for 1 year.
Arm/Group | Arm A | Arm B | Arm C (Cohort 1) | Arm C (Cohort 2) | Arm C (Cohort 3) | Arm D
All-Cause Mortality (participants affected / at risk) | 198/559 | 189/575 | 7/12 | 11/33 | 16/47 | 2/376
Serious Adverse Events (participants affected / at risk) | 82/559 | 305/575 | 6/12 | 16/33 | 30/47 | 2/376
Other Adverse Events (participants affected / at risk) | 506/559 | 529/575 | 12/12 | 32/33 | 41/47 | 7/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=559) | Arm B (N=575) | Arm C (Cohort 1) (N=12) | Arm C (Cohort 2) (N=33) | Arm C (Cohort 3) (N=47) | Arm D (N=376)
Anemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 21 | 0 | 1 | 0 | 0 — Adeers submitted
Hemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Asystole (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Cardiac arrest (Cardiac disorders) | 3 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 7 | 0 | 1 | 2 | 0 — Adeers submitted
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Heart failure (Cardiac disorders) | 4 | 15 | 0 | 1 | 2 | 0 — Adeers submitted
Left ventricular systolic dysfunction (Cardiac disorders) | 3 | 23 | 0 | 2 | 4 | 0 — Adeers submitted
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Right ventricular dysfunction (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Sinus tachycardia (Cardiac disorders) | 0 | 10 | 0 | 0 | 1 | 0 — Adeers submitted
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Ventricular arrhythmia (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Adrenal insufficiency (Endocrine disorders) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Eye disorders - Other, specify (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers submitted
Papilledema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers submitted
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 — Adeers submitted
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Anal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Colitis (Gastrointestinal disorders) | 0 | 9 | 0 | 0 | 0 | 0 — Adeers submitted
Colonic perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Diarrhea (Gastrointestinal disorders) | 0 | 9 | 0 | 1 | 0 | 0 — Adeers submitted
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 — Adeers submitted
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers submitted
Mucositis oral (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0 | 0 — Adeers submitted
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 — Adeers submitted
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 — Adeers submitted
Pancreatitis (Gastrointestinal disorders) | 0 | 8 | 0 | 0 | 1 | 0 — Adeers submitted
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Typhlitis (Gastrointestinal disorders) | 2 | 24 | 0 | 1 | 1 | 0 — Adeers submitted
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 — Adeers submitted
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Death NOS (General disorders) | 38 | 35 | 1 | 5 | 6 | 0 — Adeers submitted
Edema face (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Fever (General disorders) | 0 | 13 | 0 | 0 | 3 | 0 — Adeers submitted
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Multi-organ failure (General disorders) | 1 | 8 | 0 | 0 | 2 | 0 — Adeers submitted
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 1 | 0 — Adeers submitted
Hepatic failure (Hepatobiliary disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Allergic reaction (Immune system disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Anaphylaxis (Immune system disorders) | 0 | 5 | 0 | 0 | 0 | 0 — Adeers submitted
Immune system disorders - Other, specify (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Anorectal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Bladder infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Bronchial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Catheter related infection (Infections and infestations) | 0 | 5 | 0 | 0 | 0 | 0 — Adeers submitted
Cecal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Duodenal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Encephalitis infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Enterocolitis infectious (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Esophageal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 — Adeers submitted
Infections and infestations - Other, specify (Infections and infestations) | 2 | 13 | 0 | 2 | 0 | 0 — Adeers submitted
Lung infection (Infections and infestations) | 1 | 13 | 1 | 2 | 0 | 0 — Adeers submitted
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Mucosal infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Periorbital infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Sepsis (Infections and infestations) | 17 | 50 | 0 | 1 | 4 | 0 — Adeers submitted
Skin infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Upper respiratory infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Activated partial thromboplastin time prolonged (Investigations) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Alanine aminotransferase increased (Investigations) | 0 | 16 | 0 | 0 | 2 | 0 — Adeers submitted
Aspartate aminotransferase increased (Investigations) | 1 | 10 | 0 | 0 | 1 | 0 — Adeers submitted
Blood bilirubin increased (Investigations) | 2 | 16 | 0 | 1 | 1 | 0 — Adeers submitted
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Creatinine increased (Investigations) | 0 | 8 | 0 | 1 | 0 | 0 — Adeers submitted
Ejection fraction decreased (Investigations) | 2 | 18 | 0 | 2 | 4 | 0 — Adeers submitted
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Fibrinogen decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
GGT increased (Investigations) | 0 | 4 | 0 | 1 | 0 | 0 — Adeers submitted
Investigations - Other, specify (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 — Adeers submitted
Lipase increased (Investigations) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Lymphocyte count decreased (Investigations) | 0 | 5 | 0 | 0 | 0 | 0 — Adeers submitted
Neutrophil count decreased (Investigations) | 0 | 8 | 0 | 1 | 0 | 0 — Adeers submitted
Platelet count decreased (Investigations) | 0 | 7 | 0 | 0 | 0 | 0 — Adeers submitted
Serum amylase increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Urine output decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 — Adeers submitted
White blood cell decreased (Investigations) | 0 | 5 | 0 | 0 | 0 | 0 — Adeers submitted
Acidosis (Metabolism and nutrition disorders) | 0 | 4 | 0 | 1 | 0 | 0 — Adeers submitted
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 — Adeers submitted
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 — Adeers submitted
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 0 | 0 — Adeers submitted
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Adeers submitted
Hypernatremia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 1 | 0 — Adeers submitted
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 1 | 0 | 0 — Adeers submitted
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 8 | 0 | 0 | 0 | 0 — Adeers submitted
Hypokalemia (Metabolism and nutrition disorders) | 1 | 27 | 0 | 2 | 1 | 0 — Adeers submitted
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hyponatremia (Metabolism and nutrition disorders) | 0 | 10 | 0 | 0 | 0 | 0 — Adeers submitted
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1 | 0 | 0 — Adeers submitted
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 — Adeers submitted
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 0 | 1 — Adeers submitted
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Central nervous system necrosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Depressed level of consciousness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Dysesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Edema cerebral (Nervous system disorders) | 1 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Encephalopathy (Nervous system disorders) | 1 | 5 | 0 | 0 | 0 | 0 — Adeers submitted
Headache (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Intracranial hemorrhage (Nervous system disorders) | 2 | 3 | 0 | 0 | 0 | 1 — Adeers submitted
Leukoencephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 — Adeers submitted
Paresthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 14 | 0 | 0 | 0 | 0 — Adeers submitted
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Seizure (Nervous system disorders) | 1 | 3 | 0 | 0 | 1 | 0 — Adeers submitted
Somnolence (Nervous system disorders) | 0 | 4 | 0 | 0 | 0 | 0 — Adeers submitted
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Agitation (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 0 — Adeers submitted
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Acute kidney injury (Renal and urinary disorders) | 5 | 15 | 0 | 3 | 3 | 0 — Adeers submitted
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hematuria (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 15 | 0 | 2 | 0 | 0 — Adeers submitted
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 12 | 0 | 1 | 0 | 0 — Adeers submitted
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 0 | 1 | 0 | 0 — Adeers submitted
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 55 | 1 | 3 | 3 | 0 — Adeers submitted
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 0 | 1 | 0 | 0 — Adeers submitted
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 0 | 0 | 0 | 0 — Adeers submitted
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers submitted
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 0 | 0 | 2 | 0 — Adeers submitted
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 22 | 0 | 2 | 2 | 0 — Adeers submitted
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0 | 0 | 0 | 0 — Adeers submitted
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 — Adeers submitted
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 — Adeers submitted
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 — Adeers submitted
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Adeers submitted
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 — Adeers submitted
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 — Adeers submitted
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 10 | 1 | 2 | 3 | 0 — Adeers submitted
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers submitted
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Capillary leak syndrome (Vascular disorders) | 0 | 5 | 0 | 0 | 1 | 0 — Adeers submitted
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers submitted
Hypertension (Vascular disorders) | 0 | 10 | 0 | 1 | 1 | 0 — Adeers submitted
Hypotension (Vascular disorders) | 7 | 47 | 1 | 3 | 3 | 0 — Adeers submitted
Peripheral ischemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers submitted
Thromboembolic event (Vascular disorders) | 3 | 3 | 0 | 0 | 1 | 0 — Adeers submitted
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=559) | Arm B (N=575) | Arm C (Cohort 1) (N=12) | Arm C (Cohort 2) (N=33) | Arm C (Cohort 3) (N=47) | Arm D (N=376)
Anemia (Blood and lymphatic system disorders) | 4 | 5 | 0 | 0 | 1 | 0 — Adeers not subm
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 3 | 0 | 1 | 0 | 0 — Adeers not subm
Febrile neutropenia (Blood and lymphatic system disorders) | 212 | 175 | 6 | 8 | 12 | 2 — Adeers not subm
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Asystole (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Cardiac arrest (Cardiac disorders) | 4 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Cardiac disorders - Other, specify (Cardiac disorders) | 8 | 16 | 0 | 0 | 1 | 0 — Adeers not subm
Chest pain - cardiac (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Heart failure (Cardiac disorders) | 21 | 22 | 1 | 2 | 0 | 0 — Adeers not subm
Left ventricular systolic dysfunction (Cardiac disorders) | 30 | 28 | 1 | 1 | 0 | 0 — Adeers not subm
Pericardial effusion (Cardiac disorders) | 4 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Pulmonary valve disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Right ventricular dysfunction (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Sinus bradycardia (Cardiac disorders) | 1 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Sinus tachycardia (Cardiac disorders) | 13 | 7 | 0 | 0 | 0 | 0 — Adeers not subm
Supraventricular tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Tricuspid valve disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Ventricular arrhythmia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 — Adeers not subm
Blurred vision (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Eye disorders - Other, specify (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Periorbital edema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Vitreous hemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Abdominal pain (Gastrointestinal disorders) | 28 | 26 | 1 | 4 | 5 | 0 — Adeers not subm
Anal mucositis (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Anal pain (Gastrointestinal disorders) | 7 | 4 | 0 | 0 | 0 | 0 — Adeers not subm
Anal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Ascites (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Colitis (Gastrointestinal disorders) | 20 | 15 | 0 | 0 | 1 | 0 — Adeers not subm
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Dental caries (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Diarrhea (Gastrointestinal disorders) | 37 | 48 | 1 | 5 | 4 | 1 — Adeers not subm
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — Adeers not subm
Enterocolitis (Gastrointestinal disorders) | 2 | 8 | 0 | 0 | 0 | 0 — Adeers not subm
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Esophageal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Esophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Esophagitis (Gastrointestinal disorders) | 4 | 2 | 1 | 0 | 0 | 0 — Adeers not subm
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Gastritis (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 2 | 0 — Adeers not subm
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Ileus (Gastrointestinal disorders) | 5 | 10 | 0 | 0 | 1 | 0 — Adeers not subm
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Mucositis oral (Gastrointestinal disorders) | 115 | 92 | 4 | 10 | 11 | 0 — Adeers not subm
Nausea (Gastrointestinal disorders) | 40 | 40 | 1 | 4 | 3 | 0 — Adeers not subm
Oral hemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Oral pain (Gastrointestinal disorders) | 11 | 5 | 0 | 1 | 3 | 0 — Adeers not subm
Pancreatitis (Gastrointestinal disorders) | 2 | 5 | 0 | 2 | 1 | 0 — Adeers not subm
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Rectal mucositis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Rectal pain (Gastrointestinal disorders) | 7 | 4 | 0 | 0 | 1 | 0 — Adeers not subm
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Small intestinal mucositis (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Typhlitis (Gastrointestinal disorders) | 36 | 22 | 0 | 1 | 2 | 0 — Adeers not subm
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Vomiting (Gastrointestinal disorders) | 21 | 23 | 0 | 4 | 2 | 1 — Adeers not subm
Edema face (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Edema limbs (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Edema trunk (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Fatigue (General disorders) | 4 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Fever (General disorders) | 53 | 94 | 2 | 5 | 7 | 0 — Adeers not subm
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Localized edema (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Multi-organ failure (General disorders) | 7 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Pain (General disorders) | 13 | 13 | 1 | 1 | 4 | 0 — Adeers not subm
Cholecystitis (Hepatobiliary disorders) | 1 | 2 | 0 | 1 | 0 | 0 — Adeers not subm
Gallbladder necrosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 1 | 0 | 1 | 2 | 0 — Adeers not subm
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Allergic reaction (Immune system disorders) | 7 | 8 | 0 | 1 | 0 | 0 — Adeers not subm
Anaphylaxis (Immune system disorders) | 10 | 4 | 0 | 2 | 0 | 0 — Adeers not subm
Autoimmune disorder (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Serum sickness (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Anorectal infection (Infections and infestations) | 6 | 4 | 0 | 1 | 0 | 0 — Adeers not subm
Appendicitis (Infections and infestations) | 6 | 9 | 0 | 0 | 0 | 0 — Adeers not subm
Bladder infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Bone infection (Infections and infestations) | 5 | 1 | 1 | 0 | 0 | 0 — Adeers not subm
Bronchial infection (Infections and infestations) | 1 | 5 | 0 | 0 | 0 | 0 — Adeers not subm
Catheter related infection (Infections and infestations) | 14 | 16 | 0 | 0 | 1 | 0 — Adeers not subm
Cecal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Encephalitis infection (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 0 — Adeers not subm
Endocarditis infective (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 — Adeers not subm
Endophthalmitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Enterocolitis infectious (Infections and infestations) | 31 | 29 | 0 | 2 | 1 | 1 — Adeers not subm
Esophageal infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Gallbladder infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Gum infection (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 0 — Adeers not subm
Hepatic infection (Infections and infestations) | 4 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Hepatitis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Infections and infestations - Other, specify (Infections and infestations) | 275 | 293 | 6 | 19 | 16 | 0 — Adeers not subm
Infective myositis (Infections and infestations) | 4 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Joint infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 — Adeers not subm
Kidney infection (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Lip infection (Infections and infestations) | 0 | 4 | 1 | 0 | 2 | 0 — Adeers not subm
Lung infection (Infections and infestations) | 60 | 72 | 3 | 8 | 6 | 1 — Adeers not subm
Lymph gland infection (Infections and infestations) | 2 | 7 | 0 | 1 | 1 | 0 — Adeers not subm
Meningitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 — Adeers not subm
Mucosal infection (Infections and infestations) | 6 | 3 | 0 | 1 | 0 | 0 — Adeers not subm
Nail infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Otitis media (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 0 — Adeers not subm
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Pelvic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Penile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Periorbital infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Peritoneal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Pleural infection (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Salivary gland infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Scrotal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Sepsis (Infections and infestations) | 88 | 72 | 0 | 3 | 3 | 1 — Adeers not subm
Sinusitis (Infections and infestations) | 11 | 17 | 1 | 1 | 1 | 0 — Adeers not subm
Skin infection (Infections and infestations) | 36 | 26 | 1 | 0 | 3 | 0 — Adeers not subm
Small intestine infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Soft tissue infection (Infections and infestations) | 8 | 10 | 1 | 2 | 1 | 0 — Adeers not subm
Splenic infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Tooth infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Upper respiratory infection (Infections and infestations) | 13 | 24 | 1 | 0 | 1 | 0 — Adeers not subm
Urinary tract infection (Infections and infestations) | 18 | 20 | 0 | 1 | 1 | 0 — Adeers not subm
Vaginal infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Vulval infection (Infections and infestations) | 4 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Wound infection (Infections and infestations) | 1 | 3 | 0 | 0 | 1 | 0 — Adeers not subm
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Vascular access complication (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Venous injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Activated partial thromboplastin time prolonged (Investigations) | 6 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Alanine aminotransferase increased (Investigations) | 84 | 79 | 0 | 7 | 14 | 2 — Adeers not subm
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Aspartate aminotransferase increased (Investigations) | 56 | 63 | 0 | 5 | 7 | 1 — Adeers not subm
Blood bilirubin increased (Investigations) | 25 | 20 | 1 | 3 | 5 | 0 — Adeers not subm
CPK increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Cardiac troponin I increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Cholesterol high (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Creatinine increased (Investigations) | 1 | 10 | 1 | 0 | 1 | 0 — Adeers not subm
Ejection fraction decreased (Investigations) | 22 | 29 | 1 | 4 | 0 | 0 — Adeers not subm
Electrocardiogram QT corrected interval prolonged (Investigations) | 153 | 175 | 3 | 10 | 14 | 0 — Adeers not subm
Fibrinogen decreased (Investigations) | 1 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
GGT increased (Investigations) | 16 | 19 | 0 | 3 | 1 | 0 — Adeers not subm
INR increased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Investigations - Other, specify (Investigations) | 3 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Lipase increased (Investigations) | 10 | 9 | 0 | 1 | 0 | 0 — Adeers not subm
Neutrophil count decreased (Investigations) | 188 | 193 | 3 | 7 | 5 | 0 — Adeers not subm
Platelet count decreased (Investigations) | 4 | 7 | 0 | 0 | 0 | 0 — Adeers not subm
Serum amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Urine output decreased (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Weight gain (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Weight loss (Investigations) | 12 | 7 | 0 | 2 | 0 | 0 — Adeers not subm
White blood cell decreased (Investigations) | 2 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Acidosis (Metabolism and nutrition disorders) | 5 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Alkalosis (Metabolism and nutrition disorders) | 5 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Anorexia (Metabolism and nutrition disorders) | 123 | 130 | 5 | 7 | 11 | 0 — Adeers not subm
Dehydration (Metabolism and nutrition disorders) | 12 | 6 | 0 | 1 | 0 | 0 — Adeers not subm
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 5 | 0 | 0 | 1 | 0 — Adeers not subm
Hyperglycemia (Metabolism and nutrition disorders) | 59 | 59 | 3 | 6 | 6 | 1 — Adeers not subm
Hyperkalemia (Metabolism and nutrition disorders) | 17 | 10 | 1 | 3 | 2 | 0 — Adeers not subm
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Hypernatremia (Metabolism and nutrition disorders) | 2 | 9 | 1 | 0 | 0 | 0 — Adeers not subm
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 4 | 0 | 0 | 0 | 0 — Adeers not subm
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 | 19 | 0 | 1 | 2 | 1 — Adeers not subm
Hypocalcemia (Metabolism and nutrition disorders) | 31 | 29 | 3 | 3 | 1 | 1 — Adeers not subm
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Hypokalemia (Metabolism and nutrition disorders) | 149 | 152 | 5 | 9 | 9 | 0 — Adeers not subm
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 4 | 0 | 1 | 0 | 0 — Adeers not subm
Hyponatremia (Metabolism and nutrition disorders) | 34 | 28 | 2 | 5 | 2 | 0 — Adeers not subm
Hypophosphatemia (Metabolism and nutrition disorders) | 39 | 42 | 1 | 3 | 7 | 0 — Adeers not subm
Iron overload (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Tumor lysis syndrome (Metabolism and nutrition disorders) | 9 | 12 | 0 | 0 | 1 | 1 — Adeers not subm
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0 — Adeers not subm
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 1 | 0 | 0 | 0 — Adeers not subm
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 — Adeers not subm
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Myositis (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 1 | 0 | 0 — Adeers not subm
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 2 | 1 | 1 | 0 — Adeers not subm
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 13 | 0 | 1 | 0 | 0 — Adeers not subm
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Cognitive disturbance (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 — Adeers not subm
Depressed level of consciousness (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Headache (Nervous system disorders) | 22 | 16 | 1 | 2 | 0 | 0 — Adeers not subm
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Neuralgia (Nervous system disorders) | 0 | 3 | 0 | 1 | 0 | 0 — Adeers not subm
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Peripheral motor neuropathy (Nervous system disorders) | 4 | 11 | 0 | 0 | 1 | 0 — Adeers not subm
Peripheral sensory neuropathy (Nervous system disorders) | 15 | 29 | 1 | 2 | 2 | 0 — Adeers not subm
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Seizure (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Syncope (Nervous system disorders) | 6 | 5 | 0 | 2 | 0 | 0 — Adeers not subm
Vasovagal reaction (Nervous system disorders) | 1 | 2 | 0 | 1 | 0 | 0 — Adeers not subm
Agitation (Psychiatric disorders) | 2 | 2 | 0 | 1 | 0 | 0 — Adeers not subm
Anxiety (Psychiatric disorders) | 6 | 2 | 0 | 1 | 1 | 0 — Adeers not subm
Confusion (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Delirium (Psychiatric disorders) | 5 | 2 | 0 | 0 | 1 | 0 — Adeers not subm
Depression (Psychiatric disorders) | 4 | 0 | 0 | 1 | 1 | 0 — Adeers not subm
Hallucinations (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Insomnia (Psychiatric disorders) | 4 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Irritability (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Acute kidney injury (Renal and urinary disorders) | 7 | 9 | 0 | 1 | 0 | 0 — Adeers not subm
Cystitis noninfective (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 0 — Adeers not subm
Hematuria (Renal and urinary disorders) | 9 | 3 | 1 | 0 | 1 | 0 — Adeers not subm
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Renal calculi (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Genital edema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Menorrhagia (Reproductive system and breast disorders) | 2 | 2 | 0 | 1 | 1 | 0 — Adeers not subm
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Perineal pain (Reproductive system and breast disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Vaginal inflammation (Reproductive system and breast disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Vaginal pain (Reproductive system and breast disorders) | 1 | 2 | 0 | 0 | 1 | 0 — Adeers not subm
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 0 | 0 | 1 | 0 — Adeers not subm
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 0 | 1 | 0 | 0 — Adeers not subm
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 1 | 0 | 0 — Adeers not subm
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 1 | 1 | 0 | 0 — Adeers not subm
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 4 | 0 | 3 | 1 | 0 — Adeers not subm
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 42 | 30 | 2 | 4 | 4 | 0 — Adeers not subm
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | 1 | 0 | 0 — Adeers not subm
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 — Adeers not subm
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 1 | 0 | 1 | 0 — Adeers not subm
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 0 | 0 | 0 | 0 — Adeers not subm
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 19 | 11 | 1 | 0 | 2 | 0 — Adeers not subm
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 21 | 14 | 0 | 1 | 0 | 1 — Adeers not subm
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 0 | 0 | 2 | 0 — Adeers not subm
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — Adeers not subm
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Stridor (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Adeers not subm
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Erythroderma (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Pain of skin (Skin and subcutaneous tissue disorders) | 4 | 6 | 0 | 1 | 1 | 0 — Adeers not subm
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1 | 0 — Adeers not subm
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 2 | 0 — Adeers not subm
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 47 | 62 | 2 | 9 | 12 | 0 — Adeers not subm
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 | 2 | 0 | 0 | 0 | 0 — Adeers not subm
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 1 | 0 — Adeers not subm
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 1 | 0 | 0 — Adeers not subm
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Capillary leak syndrome (Vascular disorders) | 3 | 3 | 0 | 0 | 0 | 0 — Adeers not subm
Hematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Hypertension (Vascular disorders) | 29 | 23 | 1 | 7 | 7 | 0 — Adeers not subm
Hypotension (Vascular disorders) | 79 | 49 | 1 | 5 | 2 | 0 — Adeers not subm
Superficial thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 — Adeers not subm
Thromboembolic event (Vascular disorders) | 2 | 1 | 0 | 1 | 0 | 0 — Adeers not subm
Vascular disorders - Other, specify (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0 — Adeers not subm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT01371981/Prot_SAP_000.pdf